CLINICAL TRIAL: NCT04747613
Title: An Open Label, Multicenter Roll-over Extension Program (REP) to Characterize the Long-term Safety and Tolerability of Iptacopan (LNP023) in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Who Have Completed PNH Phase 2 and Phase3 Studies With Iptacopan
Brief Title: Long-term Safety and Tolerability of Iptacopan in Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023C12001B
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Iptacopan; Paroxysmal Nocturnal Hemoglobinuria (PNH); Hemoglobin; Anemia; LNP023
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Anemia | interventions — iptacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Iptacopan (Experimental): Participants will be receiving open label oral iptacopan 200 mg b.i.d monotherapy
  Interventions: Drug: Iptacopan

INTERVENTIONS:
Drug: Iptacopan — Taken orally b.i.d. Dosage supplied: 200 mg Dosage form: hard gelatin capsule Route of administration: oral
  Other Names: LNP023

SUMMARY:
This study is an open-label, single arm, multicenter, roll-over extension study to characterize long-term safety, tolerability and efficacy of iptacopan and to provide access to iptacopan to patients with PNH who have completed Novartis-sponsored Phase 2 or 3 studies with iptacopan

DETAILED DESCRIPTION:
The purpose of this phase 3 open-label, single arm, multicenter study is to evaluate the long-term safety, tolerability and efficacy of iptacopan in patients with PNH and to provide access to patients who have completed (without tapering down) Phase 2 and Phase 3 trials and derived benefit from iptacopan treatment.

ELIGIBILITY:
Inclusion criteria:

* Male and female participants ≥ 18 years of age with a diagnosis of PNH who have completed the treatment extension period (without tapering down) of Phase II iptacopan studies (CLNP023X2204, CLNP023X2201), Period 4 of LFG316X2201 or Phase III (CLNP023C12302 and CLNP023C12301) clinical studies at the time point of enrollment visit in this roll over extension.
* Prior vaccinations against Neisseria meningitidis, Streptococcus pneumoniae and Haemophilus influenzae infections
* Per investigator's clinical judgement benefit from continued treatment with iptacopan and has been clinically stable on iptacopan monotherapy for at least 3 months

Exclusion Criteria:

* Any comorbidity or medical condition (including but not limited to any active systemic bacterial, viral or fungal infection or malignancy) that, in the opinion of the investigator, could put the subject at increased risk or potentially confound study data.
* History of recurrent invasive infections caused by encapsulated organisms, such as Neisseria meningitidis, Streptococcus pneumoniae or Haemophilus influenzae
* History of hematopoietic stem cell transplantation

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2027-10-19 (Estimated); Study Completion 2027-10-19 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with adverse events | 60 months
  Safety evaluations including but not limited to adverse events/serious adverse events, safety laboratory parameters, vital signs, etc. through End of Study visit

SECONDARY OUTCOMES:
Proportion of participants achieving sustained hemoglobin levels ≥ 12 g/dL in the absence of red blood cell transfusions | 60 months
  Proportion of participants achieving sustained hemoglobin levels ≥ 12 g/dL in the absence of red blood cell transfusions evaluated over yearly intervals
Proportion of participants who remain free from transfusions | 60 months
  Proportion of participants who remain free from transfusions evaluated over yearly intervals
Rate of breakthrough hemolysis (BTH) | 60 months
  Rate of breakthrough hemolysis (BTH)
Proportion of participants with Major Adverse Vascular Events MAVEs | 60 months
  MAVEs (incl. thrombosis) evaluated over yearly intervals

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- United States (8):
  - City Of Hope, Duarte, California
  - USC Norris Cancer Center, Los Angeles, California
  - Univ of California Irvine (Chao Family Comprehensive Cancer Center), Orange, California
  - Lakes Research, Miami Lakes, Florida
  - Augusta University, Augusta, Georgia
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Prisma Health Upstate, Greenville, South Carolina
- Brazil (2):
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- China (2):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Tianjin
- Czechia (2):
  - Novartis Investigative Site, Ostrava, Poruba
  - Novartis Investigative Site, Brno-Bohunice
- France (5):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (6):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Riesa
  - Novartis Investigative Site, Ulm
- Italy (7):
  - Novartis Investigative Site, Ascoli Piceno, AP
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Bassano del Grappa, Vicenza
- Japan (9):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Suwa, Nagano
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Niigata
- Novartis Investigative Site, Vilnius, Lithuania
- Malaysia (2):
  - Novartis Investigative Site, Kota Kinabalu, Sabah
  - Novartis Investigative Site, Kuching, Sarawak
- Novartis Investigative Site, Nijmegen, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (3):
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
- Taiwan (2):
  - Novartis Investigative Site, Hualien City
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] DeCastro C, Sheinberg P, Han B, Vallow S, Bermann G, Dhalke M, Kumar R, Dickie G, Galipeau N, Lamoureux R, Rupinski K, Lowe C, Nieves A, de Fontbrune FS, de Latour RP. Patient-Reported Meaningful Change in Symptoms and Impacts of Paroxysmal Nocturnal Hemoglobinuria (PNH) in Three Phase III Clinical Trials of Iptacopan. Patient. 2025 Nov;18(6):699-712. doi: 10.1007/s40271-025-00755-5. Epub 2025 Jul 22. PMID 40694294